CLINICAL TRIAL: NCT06387186
Title: Open Label, Single-Arm Study of the Safety and Tolerability of a Leucine Enriched Essential Amino Acid Powder as an Add-on to a Classic Ketogenic Diet in Refractory Epilepsy
Brief Title: Leucine Enriched Essential Amino Acid Powder as an Add-on to a Classic Ketogenic Diet in Refractory Epilepsy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Elizabeth Anne Thiele (Other)
Collaborators: Ajinomoto USA, INC. (Industry); Ajinomoto Co., Inc. (Industry)
Responsible Party: Sponsor-Investigator, Elizabeth Anne Thiele, Director, Pediatric epilepsy program, Director, Herscot Center for TSC, Professor of Neurology, Harvard Medical School, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P003233
Record Dates: First submitted 2024-04-16; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Refractory Epilepsy; Drug Resistant Epilepsy
Keywords: Refractory Epilepsy; Ketogenic Diet; Leucine-Enriched Essential Amino Acid
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Leucine-Enriched Essential Amino Acid powder (LEAA) (Experimental): Leucine-Enriched Essential Amino Acid powder (LEAA) as an add-on to a classic ketogenic diet (KD)
  Interventions: Drug: Leucine-Enriched Essential Amino Acid powder

INTERVENTIONS:
Drug: Leucine-Enriched Essential Amino Acid powder — Leucine-Enriched Essential Amino Acid Powder will be orally/enterally administered by mixing in water or ketogenic formula.
  Other Names: LEAA

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of a Leucine-Enriched Essential Amino Acid (LEAA) Powder as an add-on to a classic ketogenic diet (KD) in pediatric and adult patients with refractory epilepsy.

DETAILED DESCRIPTION:
This is a single center, single-arm, open label study to evaluate the safety, tolerability, and nutritional effect of Leucine-Enriched Essential Amino Acid powder (LEAA) when added to classical KD in pediatric and adult patients whose epilepsy is insufficiently controlled on the diet. The study will enroll patients who have previously been compliant with their classical KD regimen for at least 28 days prior to enrollment and have experienced some response (≥40% reduction in seizures), but not complete response (<90% reduction in seizures) to dietary management with KD. Study duration is 84 days and will have 3 remote study visits (Baseline- Remote Visit 1, Dose Adjustment- Remote Visit 2, and Final- Remote Visit 3) and a pre-screening communication via telephone/video.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ages 2 years and up at enrollment.
2. A diagnosis of epilepsy, with at least 2 seizures per week according to the parent/guardian report to study staff and investigator medical notes if applicable. All seizure types allowed.
3. Under stable treatment with a classic ketogenic diet (KD) regimen with a KD ratio ≥ 1:1, with or without antiseizure medications (ASMs), for at least 28 days with documented, partial response (≥40% reduction in seizures), but not a complete response (<90% reduction in seizures) based on patient medical records or parental report.
4. Patient and/or parent/caregiver able and willing to follow all study procedures and successfully complete the study.

Exclusion Criteria:

1. Patients who have changed their KD regimen or antiseizure medication (ASM) or vagus nerve stimulation (VNS) within the last 28 days.
2. Allergy, sensitivity to, or inability to metabolize any component of leucine enriched essential amino acid (LEAA).
3. Those who are pregnant or breastfeeding.
4. Patients who have received an investigational drug or product or participated in a drug study within 4 weeks before the first dose of leucine enriched essential amino acid (LEAA) powder.
5. Patients who have a clinically significant condition or have had either clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to the Baseline Visit 1, other than epilepsy, that would negatively impact study participation, collection of study data, or pose a risk to the patient including liver disease.
6. Patients with history of suicidal ideation in past 6-months and suicidal behavior in past 2-years

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | Baseline, 3 weeks, 12 weeks
  Number of participants with treatment-related adverse events as reported by the trial participants.

SECONDARY OUTCOMES:
Number of participants with improved nutritional status as assessed by weight. | Baseline, 3 weeks, 12 weeks
  Nutritional status will be assessed by measuring participants' weight in kilograms.
Number of participants with improved nutritional status as assessed by body mass index (BMI). | Baseline, 3 weeks, 12 weeks
  Nutritional status will be assessed by measuring participants' weight in kilograms and height in meters to assess their body mass index (BMI).
Number of participants with improved nutritional status as assessed by serum ketone and glucose level. | At each visit and on next day
  Serum ketone and glucose level will be measure before and after intake of investigational medicine.

OTHER OUTCOMES:
Changes in seizure frequency as assessed by seizure diary. | Baseline, 3 weeks, 12 weeks
  Daily record of seizure type, duration, and frequency on seizure diary will be used to measure seizure changes.
Changes in behavior and cognitive function as assessed by a questionnaire. | Baseline, 3 weeks, 12 weeks
  Global assessment on behavior and cognitive function questionnaire will be used by study subject/parent/caregiver to assess behavior and cognitive function.
Changes in seizure severity and overall health as assessed by a questionnaire. | Baseline, 3 weeks, 12 weeks
  Global assessment on seizure severity, and overall health questionnaire will be used by clinician/dietitian and study subject/parent/caregiver to assess changes in seizure severity and overall health.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Thiele, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No